CLINICAL TRIAL: NCT01018004
Title: Prospective Randomized Trial for the Evaluation of a Theoretical Follow-Up Schedule in Cutaneous Melanoma Patients, the MELFO-Study.
Brief Title: Comparing Follow-Up Schedules in Patients With Newly Diagnosed Stage IB or Stage II Melanoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000659310; UMCG-MELFO; EU-20988
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2010-07

CONDITIONS: Melanoma (Skin)
Keywords: stage IB melanoma; stage II melanoma
MeSH Terms: conditions — Melanoma | interventions — Aftercare

INTERVENTIONS:
Other: follow-up care
Other: questionnaire administration
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Gathering information over time from follow-up visits may help doctors plan the best follow-up schedule. It is not yet known which follow-up schedule is more effective in improving patient quality of life.

PURPOSE: This randomized clinical trial is comparing follow-up schedules to see how well they work in patients with newly diagnosed stage IB or stage II melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the difference between conventional versus experimental follow-up schedules, in terms of patient well-being, expressed health-related quality of life, level of anxiety, and satisfaction with the follow-up schedule in patients with newly diagnosed stage IB or II cutaneous melanoma.
* To determine the ability of these schedules to detect recurrences and second primary melanomas in these patients.

OUTLINE: Patients are stratified according to AJCC stage (I vs II). Patients are randomized to 1 of 2 follow-up arms.

* Arm I (experimental follow-up schedule): Patients undergo a thorough history and physical examination periodically for 5 years. Patients are followed up according to the experimental schedule:

  * For stage IB disease: Patients are followed up annually for 5 years.
  * For stage IIA disease: Patients are followed up biannually for years 1 and 2 and annually for years 3, 4, and 5.
  * For stage IIB or IIC disease: Patients are followed up every 4 months during years 1 and 2, every 6 months during year 3, and annually during years 4 and 5.
* Arm II: (conventional follow-up schedule): Patients undergo a thorough history and physical examination periodically for 5 years. Patients are followed up according to the conventional schedule:

  * For all stage disease: Patients are followed up every 3 months for year 1, every 4 months for year 2, and every 6 months for years 3-5.

In both arms, patient well-being is measured at 0, 6, 12, 24, 36, 48, and 60 months after primary diagnosis, using the following questionnaires: the health-related quality of life questionnaire (RAND-36), the anxiety questionnaire (STAI version DY-1 [state] and DY-2 [trait]), the Cancer Worry Scale, and Follow-up Satisfaction questionnaire, and the self-designed specific questions regarding self-examination and follow-up satisfaction.

All patients are instructed at primary diagnosis and receive the Melanoma-Patient-Education-Package (MPEP), which consists of information on melanoma (KWF folder "melanoma") and additional instruction on self-examination. Data on type of recurrence (locoregional versus distant), the person detecting the recurrence, progression of recurrence at time of detection, the way the recurrence was detected (e.g., self-examination, accidentally, or at follow-up by physical examination or imaging) and information regarding treatment and further follow-up are collected at each follow-up visit and the outcomes are compared in both groups. Outcomes of independent questionnaires are also compared in both groups.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed newly diagnosed cutaneous melanoma

  * AJCC stage IB or II disease
* Received curative treatment
* Completed the first set of questionnaires

PATIENT CHARACTERISTICS:

* Able to speak and understand Dutch or English
* Must be able to participate in the follow-up schedule (e.g., permanently living in the Netherlands)
* No known second malignancy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2006-03; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Patient well-being expressed in 4 questionnaires

SECONDARY OUTCOMES:
Occurrence and type of recurrence (locoregional versus distant metastases) that develop
Person detecting the recurrences and the exact way of detection
Progress of recurrent disease and consequences for its treatment
Well-being of patients per group and of recurred patients

CONTACTS AND LOCATIONS:
Overall Officials: Harald J. Hoekstra, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (4):
- Netherlands (4):
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Medisch Centrum Leeuwarden - Zuid, Leeuwarden
  - Isala Klinieken - locatie Weezenlanden, Zwolle